CLINICAL TRIAL: NCT00384761
Title: Predictive Medicine Research: Investigation of Predictors of Health, Sub-clinical and Clinical Organ System Disease
Brief Title: Predictive Medicine Research
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: The Robert W. Woodruff Foundation (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Other Study IDs: IRB00024767a; PreMed 6012 (Other: Other); 1190-2005 (Other: Other)
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Atherosclerosis, Endothelial Dysfunction
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
To establish normal values by age, race, and gender of novel markers of risk in healthy subjects necessary to predict precise risk of cardiovascular disease in an individual

DETAILED DESCRIPTION:
Introduction

As a person ages their chance of developing certain diseases such as hardening of the arteries (atherosclerosis), diabetes, depression, osteoporosis and memory loss (Alzheimer's disease) increases. One of the theories that might explain why age increases the risk of developing these diseases involves a concept called oxidative stress. Oxidative stress is a process that occurs inside the cells in our body. All the cells in our body are constantly undergoing various biochemical reactions, which are important to the cell's life cycle. Byproducts of these biochemical reactions are molecules called free radicals or pro-oxidants. Pro-oxidants can be very damaging to the cell and lead to cell death. Cells also have molecules called antioxidants, which neutralize the pro-oxidants and protect the cell so it can continue functioning normally. Oxidative stress occurs when there is an imbalance in the pro-oxidants as compared with the antioxidants. Other studies have shown that diseases such as hardening of the arteries, depression, osteoporosis and Alzheimer's are associated with elevated levels of free radicals or pro-oxidants inside the cells. It is now possible to measure the levels of pro-oxidants in the cells using blood tests.

Objectives

The purpose of this study is to determine how reliable and reproducible these measurements are and also to define a "normal" value or range of values in healthy people. It is our hope that after we are able to define the normal range of values for oxidative stress we can then look at people with the aforementioned diseases and measure their levels of oxidative stress looking for a correlation between the two. If we can show a direct correlation between level of oxidative stress and these diseases we can begin trying to develop medicines that can target this area and hopefully prevent or lessen the degree of these diseases.

Tests and Evaluations

In this study we are looking for healthy participants age 30 and older who will undergo blood tests that will allow us to measure markers of oxidative stress. Participants will also undergo tests specifically designed to look for evidence of early multi-organ disease. These exams will include an evaluation of lung function (spirometry test), exercise capacity (using a stationary bike), bone density scan looking for osteoporosis, ultrasound of the artery of the neck (carotid) and artery of the arm (brachial), nerve conduction study, bio-impedance (Body fact composition) and several questionnaires to assess memory and mood. The participants require one screening visit and a follow up visit to undergo the tests.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20-90+
* Normal performance status
* LDL cholesterol level <120 mg/dl
* Fasting blood glucose <99 mg/dL
* Blood pressure <135 mmHg systolic and <85 mmHg diastolic
* Non-smoker for at least 5 years
* BMI >19 and <26; stable body weight
* Free of neurological and psychological (Axis I) disorders for at least three years.

Exclusion Criteria:

* Age <30
* Any oral antioxidants in the previous 2 weeks
* On lipid lowering medication in the past 8 weeks
* History of substance abuse
* Current cancer or history of cancer except basal cell cancer
* Any heart disease except for corrected congenital ht disease
* History of neurological disease
* History of chronic GI disorders
* History of inflammatory joint disorders
* Known endocrine disorders
* History of Chronic Pulmonary diseases e.g. COPD
* Acute illness such as infection in the previous 4 weeks
* Creatinine > 2
* Liver enzymes >1.5X normal
* Anemia (Hemoglobin < 12.5) or chronic hematological disorder
* Physical limitation and sedentary status for any reason
* LDL cholesterol > 120
* Fasting Glucose > 99
* BP >135/85 on 3 repeated measures
* Current smoker or smoker in the last 5 years
* History of depression
* Inability to give informed consent

For more information or patient referral call Johnson Pereira 404-275-0034, Rajinder Grover 404-686-7063, Muhammad Amer 404-805-4771 or Salman Sher 404-587-2667

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Individuals between ages 20-90
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2006-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Oxidative Stress | Cross Sectional

CONTACTS AND LOCATIONS:
Overall Officials: Arshed Quyyumi, MD, Principal Investigator — Emory Hospital; Muhammad Amer, MD, Study Director — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Result] Al Mheid I, Patel R, Murrow J, Morris A, Rahman A, Fike L, Kavtaradze N, Uphoff I, Hooper C, Tangpricha V, Alexander RW, Brigham K, Quyyumi AA. Vitamin D status is associated with arterial stiffness and vascular dysfunction in healthy humans. J Am Coll Cardiol. 2011 Jul 5;58(2):186-92. doi: 10.1016/j.jacc.2011.02.051. PMID 21718915
- [Result] Patel RS, Al Mheid I, Morris AA, Ahmed Y, Kavtaradze N, Ali S, Dabhadkar K, Brigham K, Hooper WC, Alexander RW, Jones DP, Quyyumi AA. Oxidative stress is associated with impaired arterial elasticity. Atherosclerosis. 2011 Sep;218(1):90-5. doi: 10.1016/j.atherosclerosis.2011.04.033. Epub 2011 May 6. PMID 21605864